CLINICAL TRIAL: NCT02652351
Title: Safety and Efficacy Study of Human Umbilical Cord-Mesenchymal Stem Cells for Hepatic Cirrhosis
Brief Title: Human Umbilical Cord-Mesenchymal Stem Cells for Hepatic Cirrhosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Hornetcorn Bio-technology Company, LTD (Industry)
Collaborators: The Second Hospital University of South China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYK-hepatic cirrhosis
Record Dates: First submitted 2016-01-07; First posted 2016-01-11 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-01

CONDITIONS: Hepatic Cirrhosis
Keywords: Stem cell; Human Umbilical Cord Mesenchymal Stem Cell; Mesenchymal Stem Cell; Hepatic Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- hUC-MSC treatment (Experimental): Patients will receive human umbilical cord mesenchymal stem cells transplantation with a 12 months follow-up.
  Interventions: Biological: Human umbilical cord mesenchymal stem cells

INTERVENTIONS:
Biological: Human umbilical cord mesenchymal stem cells — A single dose of 2×107 hUC-MSC will be implanted to patients by intravenous infusion or Hepatic artery intervention, and repeated every week for four times.
  Other Names: hUC-MSC

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of human umbilical cord mesenchymal stem cell(hUC-MSC) for Hepatic Cirrhosis.

DETAILED DESCRIPTION:
Human umbilical cord mesenchymal stem cells exhibit the potential to differentiate into mature cells typical of several tissues, which have been confirmed in in vivo and in vitro experiments. There have been few clinical reports describing umbilical cord mesenchymal stem cells for treatment of Hepatic Cirrhosis.

To investigate the effects of hUC-MSC treatment for Hepatic Cirrhosis, 20 patients with Hepatic Cirrhosis will be enrolled and receive 4 times of hUC-MSC transplantation.

ELIGIBILITY:
Inclusion Criteria:

* The patient who have signed the informed consent document;
* Clinical, radiological, or biochemical evidence of liver cirrhosis.

Exclusion Criteria:

* Pregnant women or lactating mothers;
* Patients who have received any anti-inflammatory drugs including herb-drug within 14 days;
* Patients who received any drug by intra-articular injection for treatment within 2 months prior to this enrollment;
* Patients with positive human immunodeficiency (HIV) at screening indicative of current of pass infection;
* Abnormal blood coagulation, combine other tumor or special condition;
* Patients who had participated in other clinical trials within three months prior to this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-05 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Severity of adverse events | 12 months
  According to National Cancer Institute Common Terminology Criteria for Adverse Events（NCI-CTCAE)

SECONDARY OUTCOMES:
Hepatic function | 1, 3 ,6 and 12 months
  Include AST, ALT, T-Bil and A/G.
Liver fibrosis index | 1, 3 ,6 and 12 months
  The level of Hyaluronidase,Laminin,Procollagen Ⅲ and Collagen Type IV in serum.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Chen, Professor, Principal Investigator — The second Affiliated Hospital of University of Soth China
Locations (1):
- The second Affiliated Hospital of University of Soth China, Hengyang, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided